CLINICAL TRIAL: NCT03053271
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of ATR-101 for the Treatment of Cushing's Syndrome
Brief Title: A Study of ATR-101 for the Treatment of Endogenous Cushing's Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Millendo Therapeutics US, Inc. (Industry)
Responsible Party: Sponsor
Organization: Millendo Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATR-101-301
Record Dates: First submitted 2017-02-06; First posted 2017-02-15 (Actual); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Cushing Syndrome
Keywords: Endogenous Cushing's Syndrome; ATR-101; CS
MeSH Terms: conditions — Cushing Syndrome | interventions — N-(2,6-bis(1-methylethyl)phenyl)-N'-((1-(4-(dimethylamino)phenyl)cyclopentyl)methyl)urea hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATR-101 (Experimental): During the 4-week randomized withdrawal period, eligible subjects will receive ATR-101 at the same dose level being used at the completion of the open-label dose-escalation period.
  Interventions: Drug: ATR-101
- Placebo (Placebo Comparator): During the 4-week randomized withdrawal period, eligible subjects will receive a placebo that matches the same ATR-101 dose level being used at the completion of the open-label dose-escalation period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATR-101 — During the 4-week randomized withdrawal period, subjects will be dosed for 4 weeks at the same dose level being used at the completion of the open-label dose-escalation period.
  Other Names: nevanimibe HCl
  Arms: ATR-101
Drug: Placebo — During the 4-week randomized withdrawal period, subjects will be dosed for 4 weeks with placebo that matches the same ATR-101 dose level being used at the completion of the open-label dose-escalation period.
  Arms: Placebo

SUMMARY:
This is a Phase 2 multicenter, randomized, double-blind, placebo controlled study of ATR-101 to evaluate the efficacy and safety of orally-administered ATR-101 in adults with endogenous Cushing's syndrome. Following wash-out (if needed), all eligible subjects will enter an open-label intra-subject dose-escalation period of 8 weeks' duration, followed either by a double-blind randomized withdrawal period of 4 weeks' duration (if the subject meets randomization criteria) or by an additional open label dosing period of 4 weeks' duration (if the subject does not meet randomization criteria).It is anticipated that the overall duration of the study per subject will range from approximately 16-22 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of endogenous Cushing's syndrome
* Baseline UFC 1.3 to 10 × upper limit of normal (ULN)
* If previous pituitary surgery, participants must be at least 3 months since surgery at the time of screening
* BMI between 18 and 60 kg/m2, inclusive

Exclusion Criteria:

* Pseudo-Cushing's syndrome, cyclic Cushing's syndrome or current iatrogenic Cushing's syndrome
* Candidates for surgical treatment of Cushing's syndrome, unless surgery is not anticipated to occur during the study
* Normal late night salivary cortisol or 24-hr urine free cortisol
* Radiotherapy of the pituitary within 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Findling, MD, Principal Investigator — Medical College of Wisconsin
Locations (4):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- The James Cook University Hospital, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ATR-101 (Nevanimibe HCl): Subjects received nevanimibe orally 250 mg BID for 2 weeks, then 500 mg BID for 2 weeks, then 1000 mg BID for 2-4 weeks.
Period: Overall Study
Arm/Group | ATR-101 (Nevanimibe HCl)
Started | 4
Completed | 0 (All completed the open-label dose escalation, but did not meet criteria for randomization)
Not Completed | 4
Not completed — Did not meet randomization criteria | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | ATR-101 (Nevanimibe HCl)
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3
  United Kingdom | 1
Weight [Mean (Standard Deviation); unit: kg] | 86.42 (7.755)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.79 (3.172)
24-hr Urinary Free Cortisol [Mean (Standard Deviation); unit: ug/day] — 24-hr urine samples were collected and assayed for free cortisol by liquid chromatography-tandem mass spectrometry
  ug/day | 198.84 (147.071)

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects With Either a Normal 24-hr Urinary Free Cortisol (UFC) or a Reduction in 24-hr UFC of ≥ 50% Relative to Their Baseline Value
Description: The number of subjects meeting the criterion was divided by the total number of subjects.
Time Frame: Through Day 85
Population: 4 patients were analyzed. None ("0") of them showed a normal 24-hr urinary free cortisol (UFC) or a reduction in 24-hr UFC of ≥ 50% relative to their baseline value
Measure: Count of Participants; unit: Participants
Arm/Group | ATR-101 (Nevanimibe HCl)
Number analyzed (Participants) | 4
Participants | 0
Statistical Analysis 1: Comparison: ATR-101 (Nevanimibe HCl); Test type: Other — No statistical test was done as only 4 subjects could be enrolled, none met criteria for randomization, and the study was discontinued by the Sponsor; No statistical test was done as only 4 subjects could be enrolled, none met criteria for randomization, and the study was discontinued by the Sponsor

2. Secondary Outcome: The Proportion of Subjects With a Normal 24-hr UFC
Description: The number of subjects meeting the criterion was divided by the total number of subjects.
Time Frame: Through Day 85
Population: 4 patients were analyzed. None ("0") of them showed a normal 24-hr urinary free cortisol (UFC)
Measure: Count of Participants; unit: Participants
Arm/Group | ATR-101 (Nevanimibe HCl)
Number analyzed (Participants) | 4
Participants | 0

3. Secondary Outcome: The Proportion of Subjects With a Reduction in 24-hr UFC of ≥ 50% Relative to Their Baseline Value
Description: The number of subjects meeting the criterion was divided by the total number of subjects.
Time Frame: Through Day 85
Population: 4 patients were analyzed. None ("0") of them showed a reduction in 24-hr UFC of ≥ 50% relative to their baseline value
Measure: Count of Participants; unit: Participants
Arm/Group | ATR-101 (Nevanimibe HCl)
Number analyzed (Participants) | 4
Participants | 0

4. Secondary Outcome: The Proportion of Subjects With a Normal 24-hr UFC
Description: The number of subjects meeting the criterion was divided by the total number of subjects.
Time Frame: Through Day 57 and Day 85
Population: 4 patients were analyzed at Day 57 and Day 85. None ("0") of them showed a normal 24-hr urinary free cortisol (UFC).
Measure: Count of Participants; unit: Participants
Arm/Group | ATR-101 (Nevanimibe HCl)
Number analyzed (Participants) | 4
Participants
  Day 57 | 0
  Day 85 | 0

5. Secondary Outcome: The Proportion of Subjects With a Reduction in 24-hr UFC of ≥ 50% Relative to Their Baseline Value
Description: The number of subjects meeting the criterion was divided by the total number of subjects.
Time Frame: Through Day 57 and Day 85
Population: 4 patients were analyzed at Day 57 and Day 85. None ("0") of them showed a reduction in 24-hr UFC of ≥ 50% relative to their baseline value
Measure: Count of Participants; unit: Participants
Arm/Group | ATR-101 (Nevanimibe HCl)
Number analyzed (Participants) | 4
Participants
  Day 57 | 0
  Day 85 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent until 30 days after the last dose of study drug
Arm/Group | ATR-101 (Nevanimibe HCl)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATR-101 (Nevanimibe HCl) (N=4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT03053271/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT03053271/SAP_001.pdf